CLINICAL TRIAL: NCT01333930
Title: Characterisation of Immunological Effects and Safety of Active O2 After Strenuous Exercise in Comparison With Placebo: a Double-blind, Placebo Controlled, Balanced Cross-over Study in Healthy Subjects of Both Genders With Good Fitness Level
Brief Title: Placebo Controlled Study for Characterisation of Immunological Effects and Safety of Active O2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adelholzener Alpenquellen GmbH (Industry)
Collaborators: SocraTec R&D GmbH (Other); SocraMetrics GmbH (Industry); Institut für Medizinische Diagnostik MVZ GbR (Unknown); Sport- und Rehazentrum GbR (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 1251ao10ct
Record Dates: First submitted 2011-04-08; First posted 2011-04-12 (Estimated); Last update posted 2012-05-14 (Estimated); Status verified 2012-05

CONDITIONS: Healthy
Keywords: immunological effects; Active O2; strenuous exercise; procedures; pharmacodynamic parameters; blood sampling scheme

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test product (Active O2) (Experimental)
  Interventions: Other: Active O2
- Placebo (Adelholzener Mineralwasser) (Placebo Comparator)
  Interventions: Other: Adelholzener Mineralwasser

INTERVENTIONS:
Other: Active O2 — oxygenised table water containing at least 20 mg O2 per 500 ml (15-fold higher content in comparison to placebo), further excipients: natural mineral water: carbonic acid, oxygen, sodium, potassium, magnesium, calcium, fluoride, chloride, nitrate, sulfate, hydrocarbonate (according to the summary of analysis)
  Arms: Test product (Active O2)
Other: Adelholzener Mineralwasser — natural mineral water containing the following ingredients: carbonic acid, sodium, potassium, magnesium, calcium, fluoride, chloride, nitrate, sulphate, hydrocarbonate (according to the summary of analysis)
  Arms: Placebo (Adelholzener Mineralwasser)

SUMMARY:
The aims of this study are:

* Characterisation of immunological effects of Active O2 vs. placebo after ingestion during and post standardised strenuous exercise
* Characterisation of safety and tolerability of Active O2 in comparison with placebo after ingestion during and post standardised strenuous exercise considering Adverse Events observed in the study

Moreover, the suitability of the study design shall be investigated by means of the internal pilot part, i.e. concerning applied procedures, selected pharmacodynamic parameters and blood sampling scheme.

DETAILED DESCRIPTION:
The nutritional product Active O2 (Adelholzener Alpenquellen GmbH) is a table water which contains an oxygen amount of 40 mg/l, a 15-fold higher amount compared to non-oxygenised products.

In this study the evaluation of immunological parameters which characterise the function of the immune system is planned in subjects ingesting the test product Active O2 in comparison with a placebo group. The study rationale refers to an established mechanistic hypothesis, which links gastro-intestinal hypoxia during and after strenuous exercise with an impairment of the immune system function.

During periods of exercise and physiological stress situations, the body primarily focuses on blood supply of the cardiovascular system, skeletal muscles and skin. Therefore, it is assumed that immunological effects during and after strenuous exercise are related - at least in part - to reduced blood flow in splanchnic organs which in turn leads to hypoxia induced damage of intestinal tissue, particularly the mucosal tissue, and to enhanced permeability for pathogens [1-6].

A phenomenon well described in scientific literature is related to athletes suffering from infections, particularly in the upper respiratory tract, after strenuous exercise. Significantly higher endotoxin concentrations (lipopolysaccharides) could be detected in the blood of athletes after strenuous competitions when compared to control groups [7].

In scientific studies, a decrease in the number of circulating immune cells as well as a reduced host defence function after strenuous and sustained exercise has been demonstrated in-vivo and by application of immunological in-vitro methods. Significant decreases in T-lymphocytes, T-helper cells type 1 as well as in Natural Killer cells (NK) could be shown. However, B-cells and T-helper cells type 2 are not affected in a comparable magnitude [8-10].

In one study a significant increase in regulatory T-cells (Treg) has been assessed after 45 min of swim exercise in adolescents [11]. These cells play a major role in the inhibition of effector T cell function and thus have a pronounced immunosuppressive effect. Furthermore, it has been shown that Treg-cell activity is directly linked to the occurrence of hypoxia in damaged tissues [12].

Immune responses due to exercise are complex and depend on numerous additional factors (e.g. stress hormones, reactive oxygen species) as well as on the intensity of exercise level [13-15].

Nonetheless, oxygen susceptibility of regulatory immunocompetent cells as well as integrity of the mucosal barrier function may play an important role in protection and/or modification of the immune response including the integrity of epithelial tight junctions and M-cell related transcytosis of pathogens to highly organised lymphoid structures for effective immune responses [4; 12; 16]. A strong correlation between intestinal hypoxia during strenuous exercise and the magnitude of intestinal mucosa damage has been demonstrated by plasma levels of the surrogate parameter intestinal fatty acid binding protein (I-FABP), a specific biomarker for mucosal damage in the small intestine [4; 17].

The hypothesis to be investigated in this study is that the oxygen content of Active O2 may - at least in part - compensate the hypoxic situation in the surface of the gut wall, when ingested during and after exercise. Luminal supply of oxygenated water potentially might protect mucosal tissue from ischemia related damage and could modulate immune responses. As a consequence, the overall situation of the immune system might improve. Such an effect should be reflected in the pharmacodynamic parameters determined in this study.

A first interim analysis of the previous pilot part of this study, including the results of 12 healthy subjects, revealed statistically significant differences between both treatments for leukocytes, CD8+-lymphocytes and NK cells. Significant differences in cytokine production and additional immunological parameters were not detectable in comparison of both treatments and no trends were observed which might indicate any treatment effect. Therefore, the second part of this clinical trial will be performed with a focus on the pharmacodynamic parameters from the pilot part for which statistically significant differences between treatments have been observed. However, additional inclusion of I FABP analysis is considered reasonable as this surrogate parameter specifically reflects quantifiable impairment and potential local oxygen effects on intestinal mucosa barrier function.

According to EU regulation No 1924/2006 on nutrition and health claims made on foods, nutrition producing companies must show scientific data with substantiation as a prerequisite for advertisement dealing with health related claims [17]. Thus, the clinical trial is planned to further investigate a potentially beneficial effect of Active O2 when ingested during and after exercise.

ELIGIBILITY:
Inclusion Criteria:

* sex: male/female
* age: 18 - 40 years
* body-mass index (BMI): ≥ 18 kg/m²
* good state of health
* good fitness level: determined by use of bicycle ergometer during screening phase in period pre
* written informed consent, after having been informed about benefits and potential risks of the study, as well as details of the insurance taken out to cover the subjects participating in the study

Exclusion Criteria:

* laboratory values out of normal range unless the deviation from normal is judged as not relevant for the study by the investigator
* history of or current drug or alcohol dependence
* regular intake of alcoholic food or beverages of ≥ 40 g pure ethanol for male or ≥ 20 g for female per day
* subjects who are on a diet which could affect immune response
* regular intake of caffeine containing food or beverages of ≥ 500 mg per day
* blood donation or other blood loss of more than 400 ml within the last two months prior to individual enrolment of the subject
* participation in a clinical trial/study during the last two months prior to individual enrolment of the subject
* regular treatment with any systemically available medication (except hormonal replacement therapy, e.g. hormonal contraception, thyroxine)
* pregnant or lactating women
* female subjects who do not agree to apply adequate contraceptive methods as defined in Note for Guidance on Non-Clinical Safety Studies for the Conduct of Human Clinical Trials for Pharmaceuticals (CPMP/ICH/286/95, modification), November 2000
* subjects suspected or known not to follow instructions
* subjects who are unable to understand the written and verbal instructions, in particular regarding the risks and inconveniences they will be exposed to during their participation in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2012-01; Primary Completion 2012-02 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
number of leukocytes | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of lymphocytes | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of monocytes | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of granulocytes | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of T-cells | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of NK-cells | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of CD4+ T-cells | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
number of CD8+ T-cells | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
CD4+/CD8+ Ratio | Baseline, 0h, 2h after termination of standardised exercise
  Determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.
I-FABP plasma concentration | Baseline, 0h, 2h after termination of standardised exercise
  Intestinal fatty acid binding protein; determination will be performed at the mentioned time points. Resulting values of each time point after termination of standardised exercise will be baseline corrected and results of both treatment periods will be compared. Due to design changes after the completion of an internal pilot part, both parts of the trial will be analysed and presented separately on a descriptive level (i.e. delta0, delta2). Additionally, data from parameters of both study parts will be combined using methods of meta-analysis.

SECONDARY OUTCOMES:
Absolute and relative frequency of Adverse Events (number of AEs, intensity, relationship to the test product/placebo, outcome, and seriousness as well as period and treatment) | from beginning of test product/placebo ingestion until discharge from the study (i.e. in average 1 week)
  For safety outcome measures separate analysis of each study part as well as pooled analysis including any safety data from both parts of the trial will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: Frank Donath, MD, Principal Investigator — SocraTec R&D GmbH
Locations (1):
- Sport- und Rehazentrum GbR, Erfurt, Thuringia, Germany